CLINICAL TRIAL: NCT01447602
Title: An Open Clinical Trial of IPT-A to Prevent Suicide in Depressed Adolescents With Suicidal Behavior
Brief Title: A Clinical Trial of IPT-A to Prevent Suicide in Depressed Adolescents With Suicidal Behavior
Acronym: IPT-A-CSP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6238
Record Dates: First submitted 2011-09-28; First posted 2011-10-06 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2013-04

CONDITIONS: Unipolar Depression; Dysthymia
Keywords: Major Depressive Disorder (MDD); Dysthymia; Depressive Disorder Not Otherwise Specified (DDNOS)
MeSH Terms: conditions — Depressive Disorder; Dysthymic Disorder; Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interpersonal psychotherapy (IPT-A) (Experimental): Interpersonal psychotherapy for depressed adolescents which focuses on identifying problematic relationships connected to onset or maintenance of depression and suicidal behavior. The treatment teaches skills such as communication and problem-solving to the adolescent and parents.
  Interventions: Behavioral: IPT-A

INTERVENTIONS:
Behavioral: IPT-A — Interpersonal Psychotherapy for adolescents (IPT-A) is a guideline based treatment with established efficacy as an intervention for adolescent depression

SUMMARY:
The investigators are adapting Interpersonal Psychotherapy (IPT-A) for adolescents who are referred to emergency services either for a suicide attempt or for being evaluated as high risk for suicidal behavior. The investigators will recruit 15 adolescents ages 12-19 years who present with a diagnosis of major depression, dysthymic disorder, depression disorder not otherwise specified who have a history of a suicide attempt in the past 2 months or a non-medically lethal attempt that may require psychiatric hospitalization, suicide attempt that is or report current suicidal ideation with a plan/intent, and treat them in an open clinical trial. The treatment will be conducted twice weekly for the first 8 weeks of treatment and then weekly for the remaining 12 weeks of the study. Using feedback from clinicians and participants, the investigators will make further modifications to the manual in preparation for conducting a larger controlled clinical trial.

DETAILED DESCRIPTION:
All treatment will be done on the Children's Day Unit (CDU) and the adolescent and his/her family need to agree to participate in the CDU program. The acute phase is biweekly for 8 weeks followed by weekly sessions for the remaining 12 weeks to allow for continued work on the skills and for consolidation of skills to prevent relapse. It is a total of 28 sessions in 20 weeks. There also are up to 4 additional emergency sessions that can be used to handle crises or have additional parent sessions during those 20 weeks. In addition, the child and adolescent psychiatrist will evaluate each study participant in terms of presently prescribed medication or for the need to initiate pharmacological treatment which will follow the evidence based medicine recommendations for pediatric psychopharmacology (Walkup et al., 2009). The child and adolescent psychiatrist will see each study participant weekly for monitoring of illness severity and medication management. Over the course of the 20 week treatment, the investigators will assess their diagnosis, global functioning, severity of depression, anxiety and suicidal ideation, and family factors. At each therapy session, the adolescents will be assessed for suicidal behavior by their clinician. They also will be seen every 4 weeks by an independent evaluator who will track their symptoms and functioning at weeks 4, 8, 12, 16, 20 or early termination and week 32 follow-up assessments. The open trial will allow us to determine the feasibility of recruiting depressed and suicidal youth. It also will allow us to determine the benefits of using IPT-A to treat depressed and suicidal youth.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ages 12-19 years
* English speaking adolescent
* Parent may be monolingual or bilingual in Spanish
* DSM-IV diagnosis of MDD, dysthymia, DDNOS
* Moderate impairment in functioning
* Moderate to severe depression severity
* Expressed risk for suicide or reported non-medically lethal attempt. Non-lethal attempt is defined as an attempt that did not require medical hospitalization but may require psychiatric hospitalization which often includes being in the Emergency Room for several days because there was no bed available.

Exclusion Criteria:

* Suicide attempt in the past 4 months with medical lethality that requires hospitalization which often includes being in the ER for several days because there was no bed available.
* Severe impairment in functioning
* Diagnoses of Substance abuse, Schizophrenia, bipolar disorder,Conduct disorder, primary eating disorder, Psychosis, obsessive-compulsive disorder,
* Engagement in self-injurious that requires medical treatment in the past month
* Mental retardation or severe learning disability
* Medical illness that may interfere with treatment
* Current physical or sexual abuse
* Open Administration for Children's Services (ACS) case
* Pregnancy
* Already receiving treatment for depression or have begun a medication trial for another diagnosis within the previous three months

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2011-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Score on Columbia Suicide Severity Rating Scale (C-SSRS) | Up to 42 weeks
  The C-SSRS is a scale that assesses for the presence of suicidal behavior.

SECONDARY OUTCOMES:
Change in score on Children's Depression Rating Scale (CDRS) | Week 20 and 3 month follow-up
  The CDRS is a clinician rated instrument that assesses for the presence and severity of depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Mufson, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (2):
- United States (2):
  - New York Presbyterian Hospital, New York, New York
  - New York State Psychiatric Institute, New York, New York